## Study Title: The Effect of Play on Social and Motor Skills of Children With ASD

NCT #: NCT04258254

Date: 06/01/2020

## **Statistical Plan**

Outcome measures will be obtained at the pretest and posttest. The BOT standardized motor test offers a fine-motor (precision+integration), gross motor coordination, agility and strength scores. The SIPT standardized praxis subtests provides praxis errors. t-tests or Repeated Measures ANOVA will be used to compare scores between post and pretests.

Post-intervention, the multimodal group will show improvements in the standard motor coordination variables, compared to their own baseline and compared to the control group. Specifically, we expect to see improved gross motor scores, fewer praxis errors as well as greater spontaneous verbalization in the multimodal group compared to the general movement or control group. In terms of fNIRS activation data, we expect greater multiregional activation in the multimodal group during the post-test compared to their own baseline. We expect fewer changes in activation or more localized activation in the general movement or control group.